CLINICAL TRIAL: NCT05077683
Title: Direct Oral Anticoagulants for Prevention of lEft ventRIcular Thrombus After Anterior Acute Myocardial InFarction
Brief Title: Direct Oral Anticoagulants for Prevention of lEft ventRIcular Thrombus After Anterior Acute Myocardial InFarction - APERITIF
Acronym: APERITIF
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APHP200015; 2021-001534-19 (EudraCT Number)
Record Dates: First submitted 2021-09-27; First posted 2021-10-14 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2023-07

CONDITIONS: Myocardial Infarction, Acute; Left Ventricular Thrombus
Keywords: Myocardial infarction; Left ventricular thrombus
MeSH Terms: conditions — Myocardial Infarction | interventions — Rivaroxaban

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DAPT (Active Comparator): aspirin (≤100mg per day) and P2Y12 inhibitors (i.e. clopidogrel 75mg per day or ticagrelor 90mg twice a day), as per current guidelines
  Interventions: Drug: DAPT strategy
- DAPT + Direct Oral AntiCoagulants (DOAC) (Experimental): aspirin (≤100mg per day), clopidogrel (75mg per day) or ticagrelor (90mg twice daily) and rivaroxaban 2.5mg twice daily.
  Interventions: Drug: Rivaroxaban 2.5 MG [Xarelto]; Drug: DAPT strategy

INTERVENTIONS:
Drug: Rivaroxaban 2.5 MG [Xarelto] — Experimental group: usual DAPT strategy (aspirin (≤100mg per day), clopidogrel (75mg per day) or ticagrelor (90mg twice daily)) + rivaroxaban 2.5mg twice daily.
  Arms: DAPT + Direct Oral AntiCoagulants (DOAC)
Drug: DAPT strategy — usual DAPT strategy (aspirin (≤100mg per day), clopidogrel (75mg per day) or ticagrelor (90mg twice daily)) +

SUMMARY:
APERITIF is a prospective randomized open-label, blinded end-point (PROBE) trial, nested in the ongoing the "FRENCHIE" registry, a French multicenter prospective observational study granted by "ANR-RHU Grand Emprunt", in which all consecutive patients admitted within 48 hours after symptom onset in a cardiac Intensive Care Unit (ICU) for an acute myocardial infarction (AMI) are included (NCT04050956). Among them, eligible Patients for "APERITIF" will be randomized into two groups: Dual Anti-Platelet Therapy (DAPT) alone or DAPT plus rivaroxaban 2.5mg twice daily for 4 weeks, prescribed as soon as possible after admission and completion of the initial percutaneous coronary intervention/angiography procedure.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years;
* Anterior STEMI (e.g., ST elevation above the J-point of ≥0.1 millivolt in ≥two contiguous leads or left bundle branch block) or very high-risk NSTEMI (e.g., dynamic ECG changes or ongoing chest pain or acute heart failure or hemodynamic instability independent of ECG changes or life-threatening ventricular arrhythmias) with echographic evidence of anterior wall motion abnormalities and, with a culprit lesion of the proximal or mid portion of the left anterior descending (LAD) on the coronary angiography;
* No contraindication to CMR (e.g., claustrophobia, pacemaker or defibrillator not compatible);
* Ability to provide written informed consent and willing to participate in 1-month follow-up period.
* Affiliation of social security regime.

Exclusion Criteria:

* Patients with cardiogenic shock (systolic blood pressure <90 mmHg with clinical signs of low output or patients requiring inotropic agents);
* Patients referred to surgery for coronary artery bypass grafting (CABG) or treatment of acute complications (e.g. ventricular septal rupture);
* Patients treated with fibrinolytic therapy;
* LV thrombus diagnosed before randomization using a transthoracic echocardiography;
* Active major bleeding or major surgery within the last 30 days;High bleeding risk (patients considered at increased risk of bleeding during DAPT; e.g. PRECISE-DAPT score >25; severe liver failure or Child Pugh class C);
* Known history of intracranial hemorrhagic stroke or intra-cranial aneurysm;
* Known history of peptic ulcer;
* Known stroke (any type) within the last 30 days;
* Known intolerance to aspirin, P2Y12 inhibitors, rivaroxaban and their excipients;
* Patients with presence of malignant neoplasms at high risk of bleeding
* Patients with hepatic impairment
* According to the SmPC any contraindication to rivaroxaban, aspirin, clopidogrel, ticagrelor
* Known intolerance to gadolinium chelates;
* Chronic kidney disease (creatinine clearance (ClCr) <30 mL/min);
* Indication for anticoagulation (e.g. atrial fibrillation, mechanical valves, LV thrombus…);
* Life expectancy <1 month;
* Known pregnancy at time of randomization (pregnancy test done) or breastfeeding women;
* Currently participating in another trial
* Protected adults (including individual under guardianship by court order)
* Persons deprived of their liberty by judicial or administrative decision

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 560 (Actual)
Dates: Start 2021-10-10 (Actual); Primary Completion 2023-03-10 (Actual); Study Completion 2024-02-09 (Actual)

PRIMARY OUTCOMES:
Rate of thrombus between the two arms | 1 month
  The main objective of this randomized trial is to determine whether, in anterior AMI patients (e.g., large necrosis area), the use of rivaroxaban 2.5mg twice daily in addition to DAPT (dual antiplatelet therapy) will reduce LV thrombus formation, compared with the use of DAPT alone (current practice).
  The primary endpoint is the presence of Left Ventricular (LV) thrombus at 1-month, as detected by the validated delayed enhancement (Cardiovascular Magnetic Resonance) CMR method

SECONDARY OUTCOMES:
Description of the thrombus | 1 month
  LV thrombus dimension (greatest diameter)
Rate of bleeding events | 1 month
  Rate of bleeding events using the Thrombolysis in Myocardial Infarction (TIMI) and the Bleeding Academic Research Consortium (BARC) criteria at 1 month (investigator-reported),
Rate of major adverse cardiac events (MACE) at 1 month | 1 month
  Rate of major adverse cardiac events (MACE) defined as a composite of death, non-fatal MI or stroke at 1 month
Rate of major adverse cardiac events (MACE) at 1 year | 1 year
  Rate of major adverse cardiac events (MACE) defined as a composite of death, non-fatal MI or stroke at 1-year
Rate of antithrombotic using | 1 year
  Antithrombotic drugs used in the patients with confirmed LV thrombus on CMR between 1 month and 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Etienne PUYMIRAT, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- HEGP, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Puymirat E, Soulat G, Fayol A, Mousseaux E, Montalescot G, Cayla G, Steg PG, Berard L, Rousseau A, Drouet E, Simon T, Danchin N; APERITIF study investigators. Rationale and design of the direct oral anticoagulants for prevention of left ventricular thrombus after anterior acute myocardial infarction (APERITIF) trial. Am Heart J. 2023 Dec;266:98-105. doi: 10.1016/j.ahj.2023.09.005. Epub 2023 Sep 14. PMID 37716448